CLINICAL TRIAL: NCT02202252
Title: Comparison of Single Versus Double Drains After Modified Radical Mastectomy
Brief Title: Single Versus Double Drains After Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Melih Akinci, Melih Akinci, Ankara Diskapi Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DGC-45
Record Dates: First submitted 2014-07-23; First posted 2014-07-28 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer; Mastectomy
Keywords: Patient comfort; Drains; Breast cancer; Modified radical mastectomy; Seroma
MeSH Terms: conditions — Breast Neoplasms; Seroma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single drain (Experimental): Insertion of a single drain: A negative pressure drain will be inserted below the lower flap directing to the axilla in the single drain group.
  Ultrasonography after removal of the drains: One day after removal of the drains seroma under the flaps and in the axilla will be examined by ultrasonography.
  Interventions: Procedure: Insertion of a single drain; Procedure: Ultrasonography after removal of the drains
- Double drain (Experimental): Insertion of double drains: Two negative pressure drains will be inserted into the axilla and below the lower flap in the double drains group.
  Ultrasonography after removal of the drains: One day after removal of the drains seroma under the flaps and in the axilla will be examined by ultrasonography.
  Interventions: Procedure: Insertion of double drains; Procedure: Ultrasonography after removal of the drains

INTERVENTIONS:
Procedure: Insertion of a single drain — A negative pressure drain will be inserted below the lower flap directing to the axilla.
  Arms: Single drain
Procedure: Insertion of double drains — Two drains will be inserted into the axilla and below the lower flap in the double drains group.
  Arms: Double drain
Procedure: Ultrasonography after removal of the drains — One day after removal of the drains seroma under the flaps and in the axilla will be examined by ultrasonography.

SUMMARY:
It is not known whether decreasing the number of drains used decreases patients' discomfort and duration of hospital stay without increasing seroma formation after mastectomies.

Hypothesis. Use of one drain increases patient comfort without increasing seroma formation after modified radical mastectomy (MRM) as compared to double drains.

Material and Method: Sixty patients undergoing MRM at Diskapi Yildirim Beyazit Training and Research Hospital will be randomised into single versus double drains groups. A negative pressure drain will be inserted below the lower flap directing to the axilla in the single drain group or two similar drains will be inserted into the axilla and below the lower flap in the double drains group. Drains will be removed if the output is less than 30 ml. Seroma is defined as fluid accumulation below the flaps and will be examined daily after the operation. One day after removal of the drains seroma under the flaps and in the axilla will be examined by ultrasonography. Age, body mass index smoking history, coexisting diseases of the patients duration of the hospital stay, duration of the drains in place, total drain output in the first three days after the operation and the need and frequency of aspirations due to seroma formation will be recorded. Patient comfort was measured with a comfort scale between 1-10 measuring incisional pain, pain caused by the drains, discomfort or sleep disturbances caused by the drains, The duration of the longer staying drain in the double drain group will be recorded for the duration of the drain in place parameter.

DETAILED DESCRIPTION:
Background: Seroma is one of the most common complications after mastectomies. Seroma formation results in delays in wound healing, incisional dehiscence, infections and long hospital stay. Although there are studies proving that drains do not prevent seroma formation, the use of drains for that purpose is still very common. Decreasing the number of drains used after mastectomies has been shown to decrease patients' discomfort and duration of hospital stay without increasing seroma formation.

Objective: To investigate the effects of single versus double drains on patient comfort and seroma formation after modified radical mastectomy (MRM) Material and Method: Sixty patients undergoing MRM at Diskapi Yildirim Beyazit Training and Research Hospital will be randomised into single versus double drains groups. A negative pressure drain will be inserted below the lower flap directing to the axilla in the single drain group or two similar drains will be inserted into the axilla and below the lower flap in the double drains group. Drains will be removed if the output is less than 30 ml. Seroma is defined as fluid accumulation below the flaps and will be examined daily after the operation. One day after removal of the drains seroma under the flaps and in the axilla will be examined by ultrasonography. Age, body mass index smoking history, coexisting diseases of the patients duration of the hospital stay, duration of the drains in place, total drain output in the first three days after the operation and the need and frequency of aspirations due to seroma formation will be recorded. Patient comfort was measured with a comfort scale between 1-10 measuring incisional pain, pain caused by the drains, discomfort or sleep disturbances caused by the drains, The duration of the longer staying drain in the double drain group will be recorded for the duration of the drain in place parameter. Two groups will be compared with chi-square, student's t-test or Mann-Whitney U test. P<0.005 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* Modified radical mastectomy

Exclusion Criteria:

* Distant metastasis
* Male breast cancer
* Bleeding diathesis

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Akinci M, Cetin B, Aslan S, Kulacoglu H. Factors affecting seroma formation after mastectomy with full axillary dissection. Acta Chir Belg. 2009 Jul-Aug;109(4):481-3. doi: 10.1080/00015458.2009.11680464. PMID 19803259
- [Background] Aitken DR, Minton JP. Complications associated with mastectomy. Surg Clin North Am. 1983 Dec;63(6):1331-52. doi: 10.1016/s0039-6109(16)43192-0. No abstract available. PMID 6359504
- [Background] Jain PK, Sowdi R, Anderson AD, MacFie J. Randomized clinical trial investigating the use of drains and fibrin sealant following surgery for breast cancer. Br J Surg. 2004 Jan;91(1):54-60. doi: 10.1002/bjs.4435. PMID 14716794
- [Background] Talbot ML, Magarey CJ. Reduced use of drains following axillary lymphadenectomy for breast cancer. ANZ J Surg. 2002 Jul;72(7):488-90. doi: 10.1046/j.1445-2197.2002.02456.x. PMID 12123509
- [Background] Saratzis A, Soumian S, Willetts R, Rastall S, Stonelake PS. Use of multiple drains after mastectomy is associated with more patient discomfort and longer postoperative stay. Clin Breast Cancer. 2009 Nov;9(4):243-6. doi: 10.3816/CBC.2009.n.041. PMID 19933080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period: July 2014-february 2015 Location: Dıskapi Research and training Hospital General Surgery Clinic
Groups:
- Single Drain: Insertion of a single drain: A negative pressure drain will be inserted below the lower flap directing to the axilla in the single drain group.
  Ultrasonography after removal of the drains: One day after removal of the drains seroma under the flaps and in the axilla will be examined by ultrasonography.
  Insertion of a single drain: A negative pressure drain will be inserted below the lower flap directing to the axilla.
  Ultrasonography after removal of the drains: One day after removal of the drains seroma under the flaps and in the axilla will be examined by ultrasonography.
- Double Drain: Insertion of double drains: Two negative pressure drains will be inserted into the axilla and below the lower flap in the double drains group.
  Ultrasonography after removal of the drains: One day after removal of the drains seroma under the flaps and in the axilla will be examined by ultrasonography.
  Insertion of double drains: Two drains will be inserted into the axilla and below the lower flap in the double drains group.
  Ultrasonography after removal of the drains: One day after removal of the drains seroma under the flaps and in the axilla will be examined by ultrasonography.
Period: Overall Study
Arm/Group | Single Drain | Double Drain
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Drain | Double Drain | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (11.6) | 53.9 (11.5) | 54 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patient Comfort Scale
Description: Patient comfort was measured with a comfort scale between 1-10 measuring incisional pain, pain caused by the drains, discomfort or sleep disturbances caused by the drains. 1 denotes no discomfort related to drains, 10 denotes maximum discomfort unrelieved even with nonsteroid antiinflammatory analgesics. The data will be presented by median value and range (minimum-maximum).
Time Frame: Postoperative 5 days
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Single Drain | Double Drain
Number analyzed (Participants) | 30 | 30
units on a scale | 3 [1 to 8] | 3 [1 to 9]
Statistical Analysis 1: Comparison: Single Drain vs Double Drain; Test type: Superiority or Other; p = 0.490, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Seroma Formation
Description: Seroma is defined as fluid accumulation below the flaps and will be examined daily after the operation. One day after removal of the drains seroma under the flaps and in the axilla will be examined by ultrasonography..
Time Frame: Twenty-four hours after removal of the drains up to 4 weeks
Measure: Number; unit: participants
Arm/Group | Single Drain | Double Drain
Number analyzed (Participants) | 30 | 30
participants | 18 | 10
Statistical Analysis 1: Comparison: Single Drain vs Double Drain; Test type: Superiority or Other; p = 0.035, Chi-squared

3. Other Pre Specified Outcome: Length of Hospital Stay
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 days
Measure: Median (Full Range); unit: days
Arm/Group | Single Drain | Double Drain
Number analyzed (Participants) | 30 | 30
days | 3 [2 to 7] | 3 [2 to 17]
Statistical Analysis 1: Comparison: Single Drain vs Double Drain; Test type: Superiority or Other; p = 0.819, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Groups:
- Single Drain: Insertion of a single drain: A negative pressure drain will be inserted below the lower flap directing to the axilla in the single drain group.
- Double Drain: Insertion of double drains: Two negative pressure drains will be inserted into the axilla and below the lower flap in the double drains group.
Arm/Group | Single Drain | Double Drain
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No